CLINICAL TRIAL: NCT04540523
Title: Effects of Home-based Exergaming on Preschoolers' Physical Activity and Cognition
Brief Title: Home-Based Exergaming Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project not funded
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Intervention
Record Dates: First submitted 2020-08-24; First posted 2020-09-07 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Physical Activity; Health-related Fitness; Cognition; Screen Time
Keywords: exergaming; Active video game; Home-based; preschool
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exergaming intervention group (Experimental): 30 minutes of exergaming per session and 5 sessions of exergaming play per week for a 6-month period.
  Interventions: Behavioral: Exergaming intervention group
- Traditional Physical Activity (Active Comparator): Phone consultations and workshops for parents to offer 5 times, 30 minutes per session; traditional physical activity at home for 6 months.
  Interventions: Behavioral: Traditional physical activity comparison
- Attention control group (No Intervention): Continue with usual activities at home with emailed physical activity tips.

INTERVENTIONS:
Behavioral: Exergaming intervention group — In addition to usual daily activity, the parent and child from each family will receive 3 game consoles (Wii, Kinect, and LeapTV) and various exergames (e.g., Nickelodeon Fit, Dance and Sports, Just Dance) with all necessary peripherals to play the games. Specifically, they will receive one game console and related exergames every 2 months to experience the variety of exergames and maintain interest in the games over time. Each parent will receive a booklet (established in our pilots studies) provides a standardized gameplay curriculum to play during each session, and attend training workshops at baseline and 3rd month in the PI's lab. The parent will be instructed to have the child perform exergaming at home for 30 minutes/session, 5 times per week, for 6 months. The games will be age appropriate for children 4-5-years-old. The games have been easy for children to learn and use in our pilot studies.
  Arms: Exergaming intervention group
Behavioral: Traditional physical activity comparison — Home-based behavioral (e.g., nutrition/PA) interventions for young children usually only target parent for multiple reasons. In this study, group workshop sessions will offered to parents at baseline, 3rd month and 6th month, including information concerning how to promote PA and reduce sedentary behaviors. Identical curricular contents (e.g., dance/sports) for home PA will be offered to parents at baseline and 3rd month in the PI's lab. Parents will also learn about PA and sedentary behavior and their impact on health and cognition. Meanwhile, the intervention staff will encourage parents to increase their lifestyle activity such as taking stairs instead of the elevator and housecleaning. Parents will also learn to shape their child and their PA and sedentary behaviors to attain the following goals: 2 hour or less screen time and at least 180 min. PA per day for children; and at least 150 min. moderate PA for parents per week.
  Arms: Traditional Physical Activity

SUMMARY:
This study will employ a 3-arm randomized clinical trial to determine the effects of a 6-month home-based exergaming intervention on preschoolers' physical activity, health-related fitness, cognition, and screen time, across time, at 3, 6 and 12 months, and as an exploratory outcome, will explore the moderating effects of parent involvement and physical home environment on the intervention role of exergaming across time. Briefly, a total of 330 child-parent dyads from the Twin Cities area in Minnesota will be individually randomly assigned to: 1) an exergaming intervention group (30 min. per session, 5 sessions exergaming play per week for a 6-month period); 2) a traditional PA group (phone consultations and workshops for parents to offer 5 times 30 min. PA at home for 6 months); and 3) an attention control group (continue with usual activities at home with emailed PA tips).

ELIGIBILITY:
Inclusion Criteria:

* response to an advertisement for the study;
* has only one child aged 4-5 years old in the family;
* speaks English;
* family with income within 185% of the Federal Poverty Guideline Levels determined by parents' self-report;
* has a TV with HDMI port or VGA port or video port at home
* the child has no medical conditions or physical disabilities that prohibit engagement in PA;
* physically inactive child who does not meet 120 min. PA per day;
* parental agreement to participating in the home visits and evaluations;
* lives within 20 miles of the UMN;
* family willingness to commit to 6 months of intervention and 6 months of follow-up;
* not moving out of area for the next 12 months.

Exclusion Criteria:

* children/parents from families that already own exergame(s) as these children tend to possess high experience levels with exergaming play;
* child who are physically active for more than recommended 180 min. PA per day as reported by parents.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-09-08 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity levels | 0, 3, 12 months (follow-up)
  Preschoolers' 5-day daily PA levels will be assessed using ActiGraph Link GT9X accelerometers (Pensacola, FL) at each testing cycle. The Link is lightweight and resembles a watch, and is a valid and reliable measure of PA among young children in free-living settings. Children will be instructed to wear the accelerometers on the non-dominant wrist at all times with the exception of time spent swimming for 3 weekday and 2 weekend days. In this project, activity counts will be set at 1-second epochs. Counts will be interpreted using empirically based cut points that define different PA intensities for preschoolers. Children's daily average minutes engaged in PA (MVPA and light PA) and sedentary behavior will be used as the outcome variables. Acceptable inclusion criteria for PA data will be recording of an average of 10 hours of accelerometer data per day. Compliance with wearing monitors will be facilitated according to Trost recommendations.

SECONDARY OUTCOMES:
Change in health-related fitness | 0, 3, 12 months (follow-up)
  Cardiovascular Fitness. Preschool children's cardiovascular fitness will be assessed by a modified YMCA 3-minute step test. Children will step up and down for three minutes on a 6-inch riser to a metronome beep set at 96 beats per minute (each beep corresponding to one movement of the leg with 4 beeps representing one up-down cycle). Children's heart rate will be assessed immediately before and after the conclusion of the test by the researchers via palpation of the carotid/radial artery with the child's one-minute heart rate. Children will be encouraged to do their best while performing the tests in the PAEL lab.
Change in percent body fat | 0, 3, 12 months (follow-up)
  Children's body fat percentage (bioelectrical impedance analysis) will be assessed by a TanitaBC-558 Ironman Body Composition Monitor digit weight scale.
Change in cognition | 0, 3, 12 months (follow-up)
  The computer-administered NIH Toolbox will be used to measure children's attention, inhibitory control, and cognitive flexibility. These are individually-administered tasks that require an environment that is reasonably quiet and distraction-free.
Change in screen time | 0, 3, 12 months (follow-up)
  TV allowance devices will be attached to every TV and computer in each home to track children's sedentary screen time. Exergame consoles have functions to record intervention children's playing time and thus track their active screen time. In addition, a validated screen time survey will be administered to the parents. It includes parent report of child hours spent watching TV, videos/DVD, playing video/computer games/ exergaming, surfing internet, etc. for below periods (wake-up until noon, noon until 6 pm, 6 pm until bedtime). Children's total and passive screen time will be used as the outcome variables.
Change in bodyweight | 0, 3, 12 months (follow-up)
  Children's bodyweight (in kilograms) will be assessed by aTanitaBC-558 Ironman Body Composition Monitor digit weight scale.
Change in body mass index (BMI) | 0, 3, 12 months (follow-up)
  Multiple measurements (height [cm] and weight [kg]) will be aggregated to arrive at one reported value of BMI (i.e., weight and height will be combined to report BMI in kg/m^2). To allow for growth, the BMI calculated from height and weight will be standardized using the CDC LMS method which yields BMI Z-scores for age and sex.

OTHER OUTCOMES:
Demographics and physical home environment moderators | Through study completion, an average of 1 year.
  A demographic survey, including sex, race/ethnicity, and exergaming experience, will be collected at baseline. Child's physical home environment information will be measured by a validated Home Environment Inventory. In detail, 33 items will be related to children's PA and sedentary behavior, with nearly half being assessed by direct observation (e.g., size of back yard and lawn area, number and positioning of TV and presence of other types of small screen entertainment) while the rest by parental report (e.g., family rule about TV use).
Motor skills competence covariate | 0, 3, 12 months (follow-up)
  The Test of Gross Motor Development-2 will be used to assess preschoolers' MSC. The instrument is a qualitative measure to assess the gross motor skills of children aged 3-10 years. The 5 skills tested are run, hop, jump, kick and throw. Children execute each skill twice. To evaluate skill performance, qualitative performance criteria are scored, with 1 indicating its presence and 0 its absence. If a skill is assessed using three performance criteria, the raw scores can therefore vary between 0-6. The highest raw total subtest score for the locomotor as well as the object control skills. Higher scores mean a better outcome.
Perceived competence covariate | 0, 3, 12 months (follow-up)
  To examine children's perceived competence, the validated Pictorial Scale of Perceived Competence and Social Acceptance (PSPCSA)106 for preschool children will be used. In detail, the subscale of perceived physical competence will be assessed. A sample of the survey is provided in Appendix 1. Enjoyment. A modified Physical Activity Enjoyment Scale will be used to assess preschool children's enjoyment toward physical activity. This scale will use similar pictorial scale as the PSPCSA and has 4 levels for the children to choose for each item. It has shown acceptable validity for use with the preschool children. The scales will be individually administered at baseline in the PI's lab to protect the privacy of the child. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota - Twin Cities, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No